CLINICAL TRIAL: NCT02780557
Title: A Randomised Control Trial to Test the Effect of Parent Contingent Talk During Shared Book Reading on Infant Language Learning.
Brief Title: How Parents Can Help Babies Learn to Talk With Picture Books.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Danielle Matthews, Reader in Cognitive Development, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R/139470-11-1-INFANCY
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Language Development
Keywords: Vocabulary; Book reading; Infancy; Parenting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingent Reading Intervention (Experimental)
  Interventions: Behavioral: Contingent Reading Intervention
- Book Provision Control (Other)
  Interventions: Behavioral: Book Provision Control

INTERVENTIONS:
Behavioral: Contingent Reading Intervention — Caregivers will be provided with 6 picture books. They will be trained to use contingent talk when looking at picture books with their infants. They will be asked to spend 10 mintues each day engaging in contingent talk while looking at picture books. The intervention will run for 4 months. Parents will be asked to keep a daily reading diary.
  Arms: Contingent Reading Intervention
Behavioral: Book Provision Control — Caregivers will be provided with 6 picture books. They will not be trained to read with their child. They will receive information from other sources (e.g. health visitors and Book Start schemes) as normal.
  Arms: Book Provision Control

SUMMARY:
The aim of this project is to test whether giving parents advice about book reading is effective in promoting language learning for infants from a range of socio-economic backgrounds.

DETAILED DESCRIPTION:
Children from disadvantaged families tend to have limited language skills compared to their advantaged peers. While many factors contribute to language ability, two aspects of the early caregiving environment are known to be correlated with child language outcomes 1) caregiver-child book reading and 2) caregiver contingent talk. Contingent talk refers to a style of communication whereby the caregiver talks about what is in their infant's current focus of attention. This style of talking can be facilitated when parents read books with their babies. The aim of this research is to establish whether asking parents to engage in contingent talk in the context of book reading promotes vocabulary learning. This study will compare the effects of an intervention to promote contingent talk against a control where parents are given books but not given any training in how to read them in a contingent manner. The study will include children from socio-economically advantaged and disadvantaged families.

ELIGIBILITY:
Inclusion Criteria:

Infants must be:

* first born and singletons
* full term (i.e. born no more than 3 weeks prematurely)
* with birth weight over 2.5 kg.

Primary caregivers must:

* work less than 24 hours per week (i.e., be the caregiver the child spends most time with)
* be raising their child as monolingual English speakers.

Exclusion criteria:

Neither caregivers nor infants must have any significant known physical, mental or learning disability.

Ages: 11 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Change in infant expressive vocabulary | Baseline: 11 months, outcome: 15 months
  Parents will complete a standardised assessment of vocabulary, the MacArthur-Bates Communicative Development Inventory (CDI).

SECONDARY OUTCOMES:
Change in caregiver reported frequency of reading | Baseline: 11 months, outcome: 15 months
  Parents will complete a questionnaire about how frequently they read with their child.
Infant Real Time Language Understanding: Accuracy | 15 months
  Infants' real-time comprehension of familiar words will be assessed at 15 months using the looking-while-listening (LWL) procedure (Fernald et al., 2008). Infants will sit in front of a computer screen with a picture on either side of it (e.g., a bottle and a shoe). We will measure the accuracy with which they look to the correct picture upon hearing a word that describes it.
Infant Real Time Language Understanding: Reaction Time | 15 months
  Infants' real-time comprehension of familiar words will be assessed at 15 months using the looking-while-listening (LWL) procedure (Fernald et al., 2008). We will measure the time it takes the child to look from a distractor to the target.

OTHER OUTCOMES:
Change in caregiver contingent talk while book reading | Baseline: 11 months, outcome: 15 months
  Video recordings of dyads reading books will be analysed for quantity of caregiver contingent talk.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Matthews, PhD, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
With participants' permission, IPD will be archived in accordance with the guidelines of the University of Sheffield, the UK Data Archive and the ESRC's Research Data Policy.